CLINICAL TRIAL: NCT04965545
Title: Role for Biochemical Assays and Kayser-Fleischer Rings in Diagnosis of Wilson Disease
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: WD-Biochemical assays
Record Dates: First submitted 2021-07-05; First posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Wilson Disease
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — This study was approved by the ethics committees of the local hospitals. After obtaining informed consent from the affected individuals or legal guardians, genetic DNA were collected and reserved.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Wilson's disease cohort: Patients were clinically diagnosed according to the Leipzig Score and included in the study when they were confirmed to carry ATP7B pathogenic variants in 2 different alleles.
  Interventions: Dietary Supplement: low copper diet

INTERVENTIONS:
Dietary Supplement: low copper diet — All patients with wilson disease should receive low copper diet

SUMMARY:
The investigators aimed to identify factors associated with symptoms and features of Wilson disease from a large cohort during long-term follow-up

DETAILED DESCRIPTION:
Wilson disease is an autosomal recessive disorder that impairs copper homeostasis and is caused by homozygous or compound heterozygous mutations in ATP7B, which encodes a copper-transporting P-type ATPase. Patients have variable clinical manifestations and laboratory test results, resulting in diagnostic dilemmas. Therefore, the investigators aimed to identify factors associated with symptoms and features of Wilson disease, thereby give timely diagnosis for patients.

ELIGIBILITY:
Inclusion Criteria:

* genetically diagnosed patients with wilson disease

Exclusion Criteria:

* Deny follow-up

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with wilson disease
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2004-01-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Serum ceruloplasmin | From 2004 through 2030
  Serum ceruloplasmin levels were collected among patients with wilson disease. After confirming a non-Gaussian distribution, the reference range of serum ceruloplasmin level was determined.
Urinary Copper Excretion | From 2004 through 2030
  The measurement of 24-hour urine copper excretions were collected and measured.
Kayser-Fleischer Rings | From 2004 through 2030
  The presence of Kayser-Fleischer Rings among patients with wilson disease were confirmed via slit lamp.
Brain Magnetic Resonance Imaging | From 2004 through 2030
  Brain Magnetic Resonance Imaging of all patients were collected and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Ying Wu, Principal Investigator — Second Affiliated Hospital, Zhejiang University School of Medicine
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No